CLINICAL TRIAL: NCT03170947
Title: Effects of Insoles in Patients With Rheumatoid Arthritis Through Measurement of Quality of Life and Physical Activity: Randomized Controlled Trial.
Brief Title: Effects of Insoles in Patients With Rheumatoid Arthritis: Randomized Controlled Trial.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Gabriel Gijon-Nogueron, Principal Investigator, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNIMalaga
Record Dates: First submitted 2017-05-26; First posted 2017-05-31 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Foot; Insoles; Quality of life; Physical Activity
MeSH Terms: conditions — Arthritis, Rheumatoid; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Custom insoles (Experimental): Custom insoles will make with CAD-CAM using a laser scanning and casting for its construction. Custom insoles will make with direct adaptation technique (TAD) being of pvc resin.
  Interventions: Device: Custom Insoles
- Standardized insoles (Active Comparator): Standardized insoles will be done by Ethylene-vinyl acetate (EVA) material.
  Interventions: Device: Standardized insoles

INTERVENTIONS:
Device: Custom Insoles — Custom insoles will make with CAD-CAM using a laser scanning and casting for its construction. All this needs the assistance of a computer. From the digital image of a positive of the limb in foam the insole will be obtained.
  Custom insoles make with direct adaptation technique (TAD) being of pvc resin. Once the resins are cut and with a temperature of 90º, they will be adapted to the foot (which will be protected with a sock) of the patient with the help of a vacuum. To this technique subtalar joint will be in a neutral position and metatarsal joints will be aligned.
  Arms: Custom insoles
Device: Standardized insoles — Standardized insoles were done by EVA material with shore of 18 and 180 kg/cm3 and manufactured, with an extension of 3/4. It was in contact with heel and plantar arch.
  Arms: Standardized insoles

SUMMARY:
Deformity and foot pain is nearly omnipresent (90%) in rheumatoid arthritis (RA), due to the interaction between inflammation and abnormal biomechanical. These cause instability in the hindfoot, which cause deformity of the forefoot, and they cause more pressure on the plantar forefoot and more pain during daily activities. Non-pharmacological interventions (insole, footwear) have an important role, reducing pain and disability, increasing the effectiveness and improving daily activities.

DETAILED DESCRIPTION:
Randomized double-blind clinical trial. Two samples of patients will be taken: the control group, which will consist of patients with rheumatoid arthritis and standardized insoles, and other group, which will consist of patients with rheumatoid arthritis and insoles made with direct adaptation technique (TAD) and patients with rheumatoid arthritis and insoles made with an scanner (CAD-CAM). The variables that the investigators will measure are: age, sex, study level, current occupation, rheumatoid arthritis evolution time, quality of life and physical function, pain and health level and general function of the foot. The investigators will use: an accelerometer, and questionnaires: Foot and Ankle Ability Measures (FAAM), Manchester foot pain and disability index (MFPDI), Medical outcomes study short form-36 (SF-36) y Foot Function Index (FFI). This study will analyze patients in the Universities of Malaga and Salford for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years of age
* Early RA
* To meet the criteria of American College of Rheumatology
* History of bilateral subtalar and/or ankle and/or talonavicular pain
* Informed consent
* Normal range of motions at the ankle, subtalar, and midtarsal joints.

Exclusion Criteria:

* Concomitant musculoskeletal disease
* Central or peripheral nervous system disease
* Endocrine disorders, especially diabetes mellitus with a level of insufficient foot sensitivity
* Patients with a history of orthopedic foot surgery
* Those currently using foot orthoses.
* Patients with foot trauma in the last 6 months previous to the study
* Vascular diseases affecting the foot, active synovitis and edema.
* Normal daily walking aids will be not permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2022-01-21 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Active graph (bracelet) at 3 months | one week, one month and three months
  This outcome will be measured with an activity monitor, accelerometer

SECONDARY OUTCOMES:
Change from Baseline quality of life at 3 months | one week, one month and three months
  This outcome will be measured with a self-reported questionnaire (SF-36)
Change from Baseline foot function 3 months | one week, one month and three months
  This outcome will be measured with a self-reported questionnaire (foot function index)
Change from Baseline pain intensity at 3 months | one week, one month and three months
  This outcome will be measured with a self-reported questionnaire (Manchester foot pain and disability index)
Change from Baseline physical activity at 3 months | one week, one month and three months
  This outcome will be measured with a self-reported questionnaire (foot and ankle ability measure)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Gijon Nogueron, PhD, Principal Investigator — University of Malaga
Locations (1):
- University of Malaga, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramos-Petersen L, Nester CJ, Ortega-Avila AB, Skidmore S, Gijon-Nogueron G. A qualitative study exploring the experiences and perceptions of patients with rheumatoid arthritis before and after wearing foot orthoses for 6 months. Health Soc Care Community. 2021 May;29(3):829-836. doi: 10.1111/hsc.13316. Epub 2021 Feb 9. PMID 33560583
- [Derived] Ramos-Petersen L, Nester CJ, Gijon-Nogueron G, Ortega-Avila AB. Foot orthoses for people with rheumatoid arthritis, involving quantitative and qualitative outcomes: protocol for a randomised controlled trial. BMJ Open. 2020 Jul 19;10(7):e036433. doi: 10.1136/bmjopen-2019-036433. PMID 32690521